CLINICAL TRIAL: NCT01905566
Title: Comparison of Clopidogrel Versus Ticagrelor Therapy for Atherosclerotic Plaque Inflammation: Serial FDG PET/CT Imaging Study of Carotid Artery and Ascending Aorta
Brief Title: Comparison of Clopidogrel Versus Ticagrelor Therapy for Atherosclerotic Plaque Inflammation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CHEOL WHAN LEE, M.D., Ph.D (Other)
Collaborators: AstraZeneca (Industry); CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, CHEOL WHAN LEE, M.D., Ph.D, MD, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMCCV2012-02
Record Dates: First submitted 2013-07-19; First posted 2013-07-23 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-02

CONDITIONS: Plaque, Atherosclerotic
Keywords: Plaque, Atherosclerotic; clopidogrel; ticagrelor; Fluorodeoxyglucose F18; Positron-Emission Tomography and Computed Tomography
MeSH Terms: conditions — Plaque, Atherosclerotic | interventions — Clopidogrel; Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clopidogrel (Active Comparator): clopidogrel: 75mg once a day
  Interventions: Drug: Clopidogrel
- Ticagrelor (Experimental): ticagrelor: 90mg twice a day
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Clopidogrel — 75mg once a day
  Arms: Clopidogrel
Drug: Ticagrelor — 90mg twice a day
  Arms: Ticagrelor

SUMMARY:
Objectives: To compare the effects of clopidogrel versus ticagrelor on atherosclerotic plaque inflammation using serial FDG PET/CT imaging of carotid artery and ascending aorta.

Hypothesis: Thrombosis and inflammation are tightly linked rather than separate entities. Therefore, P2Y12 receptor inhibitors may have an anti-ischemic effect by inhibiting plaque inflammation, and ticagrelor may be superior in efficacy to clopidogrel.

ELIGIBILITY:
Inclusion Criteria:

* Men or Women at least 18 years of age inclusive
* Patients with acute coronary syndromes (unstable angina pectoris Braunwald class IB, IC, IIB, IIC, IIIB, IIIC, NSTEMI or STEMI)
* FDG PET/CT shows at least 1 hot uptakes at carotid and or ascending aorta
* The patient or guardian agrees to the study protocol and the schedule of clinical and FDG PET/CT follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethical Committee of the respective clinical site.

Exclusion Criteria:

* Patients treated with carotid endarterectomy or stent placement
* Chronic disease requiring treatment with oral, intravenous, or intra-articular corticosteroids (use of topical, inhaled, or nasal corticosteroids is permissible).
* Untreated hyperthyroidism, or hypothyroidism
* Any clinically significant abnormality identified at the screening visit, physical examination, laboratory tests, or electrocardiogram which, in the judgment of the Investigator, would preclude safe completion of the study.
* Evidence of congestive heart failure, or left ventricular ejection fraction < 40%.
* Significant renal disease manifested by serum creatinine > 2.0mg/dL, or creatinine clearance of < 40 ml/min (by Cockcroft-Gault method).
* Hepatic disease or biliary tract obstruction, or significant hepatic enzyme elevation (ALT or AST > 3 times upper limit of normal).
* History of adult asthma manifested by bronchospasm in the past 6 months, or currently taking regular anti-asthmatic medication(s).
* Unwillingness or inability to comply with the procedures described in this protocol.
* Patient's pregnant or breast-feeding or child-bearing potential.
* Type I Diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-09; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
change (follow-up minus baseline) in standardized FDG uptake value within the regions of interest | 6months
  Analyses of FDG activity will be quantified on common carotid arteries and ascending aorta of the aortic arch. Primary endpoint is change (follow-up minus baseline) in standardized FDG uptake value within the regions of interest, known as a target-to-background ratio(blood-normalized standardized uptake value).

SECONDARY OUTCOMES:
Serial changes of high-sensitivity C-reactive protein | 6months
Serial changes of lipid battery | 6months
  lipid battery (total cholesterol, triglyceride, HDL-cholesterol, LDL-cholesterol).

CONTACTS AND LOCATIONS:
Overall Officials: Cheol-whan Lee, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea